CLINICAL TRIAL: NCT05588427
Title: Effect of Ketone Ester Supplementation on Hypoxic Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Chiel Poffé, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S66320
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Ketosis; Hypoxia
Keywords: Acute Mountain Sickness; Sleep; Cognitive Decline
MeSH Terms: conditions — Ketosis; Hypoxia; Altitude Sickness; Cognitive Dysfunction | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: 1 session with ketone ester supplementation and 1 session with taste and viscosity matched placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone group (Experimental): Ketone esters will be provided
  Interventions: Dietary Supplement: Ketone ester
- Placebo group (Placebo Comparator): Ketone placebo will be provided
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone ester — A total of 240g ketone ester supplementation will be provided in one of the 28h experimental sessions in order to establish intermittent exogenous ketosis. Sucralose (5% w/w) is added to the ketone ester (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
  Arms: Ketone group
Dietary Supplement: Placebo — Water, 5% sucralose (w/w), octaacetate (1 mM)
  Arms: Placebo group

SUMMARY:
This WP specifically aims to elucidate the effects of IEK on hypoxic tolerance and the development and severity of AMS symptoms, blood and tissue oxygenation status, as well as sleep quality during an episode of acute exposure to severe hypoxia.

DETAILED DESCRIPTION:
Acute altitude exposure impairs exercise tolerance and performance, decreases the rate of maximal oxygen uptake (V̇O2max), cognitive function and sleep quality, and often also induces symptoms of acute mountain sickness (AMS). Previous studies have clearly indicated that ketone bodies exert a neuroprotective effect under hypoxic-ischemic conditions as well as improve hypoxic tolerance in rodents. In support of these earlier observations, recent pilot experiments in young volunteers in our laboratory provide proof of concept that IEK can attenuate oxygen desaturation during exercise in hypoxia. Therefore, given that impaired exercise tolerance in hypoxia is primarily due to impaired oxidative energy production in active tissues (brain and muscle), we hypothesize that IEK can increase blood and tissue (muscle and brain) oxygenation status in hypoxia and thereby enhance global hypoxic tolerance, as well as improve exercise tolerance and endurance exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 35 years old
* Body Mass Index (BMI) between 18 and 25
* Physically fit and regularly involved in physical activity (2-5 exercise sessions of > 30min per week)
* Good health status confirmed by a medical screening
* Non smoking
* Normal sleep pattern as assessed by the Pittsburgh Sleep Quality Index (PSQI, appendix 2)

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication for hypoxic exposure and/or to perform high-intensity exercise
* Intake of any medication or nutritional supplement that is known to affect exercise, performance or sleep
* Intake of analgesics, anti-inflammatory agents, or supplementary anti-oxidants, from 2 weeks prior to the start of the study.
* Recent residence or training under hypoxia; more than 7 days exposure to altitude > 1500m during a period of 3 months preceding the study.
* Night-shifts or travel across time zones in the month preceding the study
* Blood donation within 3 months prior to the start of the study
* Smoking
* More than 3 alcoholic beverages per day
* Involvement in elite athletic training at a semi-professional or professional level
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in incidence of acute mountain sickness symptoms | Hour 0 - Hour 4 - Hour 10 - Hour 24 - Hour 28
  Scored by Lake Louise Scoring system
Change in oxygenation status of brain, blood, muscle | Hour 1 - Hour 4 - Hour 10 - Hour 24 - Hour 28
  Measured by NIRS, pulse oximetry, blood samples
Change in cerebral blood flow | Hour 1 - Hour 4 - Hour 10 - Hour 24 - Hour 28
  Measured using duplex ultrasound
Time in hypoxia | From start of hypoxic exposure until subjects are too sick to comply to (supplementation) protocol or until end of protocol, up to 29 hours
  Total time that subjects were able to comply to the experimental protocol and supplementation protocol

SECONDARY OUTCOMES:
Sleep quality | Throughout the entire duration of the night, up to 9 hours after individual bedtime
  Measured using polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Chiel Poffé, Dr., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No